CLINICAL TRIAL: NCT04507009
Title: Clinical Investigation of the Efficacy of CGF (Concentrated Growth Factor) and Ozone in the Treatment of Alveolar Osteitis
Brief Title: Clinical Investigation of the Efficacy of CGF and Ozone in the Treatment of Alveolar Osteitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dr. Damla Torul, Associate Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-2005
Record Dates: First submitted 2020-08-04; First posted 2020-08-10 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Alveolar Osteitis
Keywords: Alveolitis; Dry socket; Ozone; CGF
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Traditional treatment group which alvogyl applied to the socket after irrigation
  Interventions: Other: Traditional treatment
- Ozone (Experimental): Ozone group which Ozone (O3) applied after irrigation of the socket
  Interventions: Device: Ozone
- CGF +Ozone (Experimental): CGF + Ozone group which concentrated growth factor (CGF) after Ozone (O3) applied followed by irrigation of the socket.
  Interventions: Device: Ozone; Other: CGF

INTERVENTIONS:
Device: Ozone — topical gaseous ozone application
  Arms: CGF +Ozone; Ozone
Other: CGF — concentrated growth factor (CGF) application
  Arms: CGF +Ozone
Other: Traditional treatment — Alvogyl application
  Arms: Control

SUMMARY:
The aim of this study is to investigate the efficacy of CGF and Ozone in the treatment of alveolitis and to develop a new treatment protocol that can enable a quick and effective solution of this clinical problem, which significantly affects patients' comfort of life.

DETAILED DESCRIPTION:
In the present study, 60 healthy patients > 18 years old and have alveolitis, will included. 60 patient will divided randomly into three groups as Control, Ozone and Ozone+CGF. After irrigation of the sockets alvogyl, ozone and ozone+CGF will applied to the sockets respectively. Post operative pain, will measured at 1st to 7th days. Post operative infection, and granulation tissue will measured at 1st, 3rd and 7th days. Oral hygiene will evaluated at first visit. Quality of life will evaluated at 7th day.

ELIGIBILITY:
Inclusion Criteria:

Patients who have one or more of the following in addition to severe pain, which occur within and around the socket 1-3 days after extraction and do not decrease with pain killers;

* With a partially or completely disintegrated blood clot in the socket
* With exposed bone that gives a dark gray appearance
* With bad odor

Exclusion Criteria:

* Who does not want to be volunteer for the study,
* Smokers,
* During pregnancy or lactation,
* Has a chronic systemic disorder that will affect recovery,
* Has hematological disorder
* Cooperation cannot be established,
* Previously received radiotherapy or chemotherapy,
* Patients using oral contraceptives

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in post-operative pain assessed: visual analog (VAS) scale | 6th and 24th hour, 2nd day, 3rd day, 4th day, 5th day, 6th day and 7th day
  For the evaluation of the pain, the visual analog scale (VAS) will be used to express the absence of pain in the initial part on a straight line (0) and the end part to express the unbearable pain (10).
  0 (no pain)--------------------------------------------------------------------------------10 (unbearable pain) Higher values of the scale represent worse outcome.

SECONDARY OUTCOMES:
Granulation tissue health | postoperative 1st, 3rd, 7th days
  Granulation tissue formation in the area after treatment will be evaluated clinically. Granulation tissue will be scored as healthy (pink color and no bleeding on probing) and unhealthy granulation tissue (dark red in color and usually bleeding on probing).
Inflamation severity | postoperative 1st, 3rd, 7th days
  The severity of inflammation will be assessed using the gingival index; From values 0 to 3; 0.Normal gingiva
  1. Slight inflammation-slight discoloration, mild edema. no probing on bleeding,
  2. Moderate inflammation - redness, edema. bleeding on probing,
  3. Severe inflammation-marked redness and edema, ulceration and tendency to spontaneous bleeding
Change in the quality of postoperative life after the procedures performed | postoperative 7th day
  The evaluation of the change in postoperative quality of life will be done with a scale of post-operative symptom severity (PoSSe) consisting of 15-item questionnaire in which the effect of operation on eating, speech, sensation, appearance, pain, disease and daily activities is evaluated. This questionnaire was divided into subscales corresponding to seven main adverse effects, and for each possible answer there was a score ranging from 0 to a variable number. For total possible answer there was a score ranging from 0 to a 97.9. Higher values of the scale represent worse outcome.

OTHER OUTCOMES:
Oral hygiene degree | Evaluation of the oral hygiene before operation
  Oral hygiene of the patient will be evaluated in 3 groups as poor, moderate and good.
  * Good
    * Patients with a low incidence of active caries,
    * Patients with no bleeding and non-inflamed gums, as well as no plaque, calculus, and gingival pocket formation.
  * Bad
    * Patients with periodontitis, inflamed gums, bleeding on probing, pocket formation,calculus
    * Patients with active caries.
  * Moderate
    * Patients other than these two groups will be evaluated as moderate.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Torul, DDS PhD, Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD can share with other researchers on demand